CLINICAL TRIAL: NCT05962554
Title: IJobs - an Internet Intervention for the Unemployed: a Randomized Controlled Trial
Brief Title: IJobs - an Internet Intervention for the Unemployed
Acronym: iJobs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCT iJobs
Record Dates: First submitted 2023-06-19; First posted 2023-07-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-11

CONDITIONS: Unemployment
Keywords: iJobs

STUDY DESIGN:
Intervention Model Description: The two independent groups (intervention vs. waiting list control group) will be crossed with three measurement times (i.e., baseline, post-intervention, and 1-month follow-up). Hence, the design will be a 2 (intervention vs. control) X 3 (baseline, post-intervention, and 1-month follow-up) factorial design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The group that will be first randomly allocated to iJobs.
  Interventions: Behavioral: iJobs
- Waiting list control group (Experimental): This group will receive the intervention 2-weeks after the intervention group finishes it.
  Interventions: Behavioral: iJobs

INTERVENTIONS:
Behavioral: iJobs — iJobs is a 2-week intervention consisting of 5 modules focusing on discovering job skills, job search strategies, preparing effective resumes, exercising different types of interviews, and overcoming setbacks in the job search process. This is an adaptation of the JOBS program.

SUMMARY:
The current study aims to test the efficacy of iJobs, an online intervention for the unemployed. iJobs is an online adaptation of the JOBS program.

DETAILED DESCRIPTION:
The current study is a two-arm randomized controlled trial that will test the efficacy of iJobs (a web-based adaptation of the JOBS program) against a waiting list control group. Participants from the control group will be enrolled in iJobs 2 weeks after the experimental group finishes the program. iJobs is a 2-week intervention consisting of 5 modules focusing on discovering job skills, job search strategies, preparing effective resumes, exercising different types of interviews, and overcoming setbacks in the job search process. iJobs was previously tested in a feasibility and acceptability trial.

ELIGIBILITY:
Inclusion Criteria:

* Unemployed and looking for a job
* Work as volunteers and are looking for a paid job
* Have a PC or laptop and basic digital competencies

Exclusion Criteria:

* They don't have internet access and are not available during the two weeks of the program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Participants' self-efficacy regarding the job search process | Change from baseline to post-intervention and follow-up (approximately 2 weeks and 6 weeks)
  The Job Search Self-Efficacy Scale (20-item) measures participants' perception of their ability to gain employment. The minimum score is 20 and the maximum is 100. A higher score means a better outcome (increased job search self-efficacy).
Participants' job search intensity and effort | Change from baseline to post-intervention and follow-up (approximately 2 weeks and 6 weeks)
  The investigators will use a version of Blau's Job-search behaviors scale adapted to the contemporary context and Romanian population. The scale measures participants' involvement in job search activities in terms of frequency and intensity. The minimum score is 16 and the maximum is 80. A higher score means a better outcome (increased job search behavior effort).
The quality of participants' job search behaviors | Change from baseline to post-intervention and follow-up (approximately 2 weeks and 6 weeks)
  The Job search quality scale has 20 items and measures the quality in which the job search behaviors are performed. The minimum score is 20 and the maximum is 100. A higher score means a better outcome (increased job search quality).

SECONDARY OUTCOMES:
Participants' ability to deal with setbacks in the job search process | Change from baseline to post-intervention (approximately 2 weeks)
  Inoculation against setbacks (i.e., participants' ability to deal with setbacks) will be measured using 2 items retrieved from previous studies. The minimum score is 2 and the maximum is 10. A higher score means a better outcome (presence of inoculation against setbacks).
Participants' overall self-esteem | Change from baseline to post-intervention (approximately 2 weeks)
  Rosenberg's Self Esteem Scale measures global self-worth by measuring both positive and negative feelings about the self using 10 items. The minimum score of Rosenberg's Self Esteem Scale is 10 and the highest one is 40. A higher score means a better outcome.
Participants' anxiety regarding their future career | Change from baseline to post-intervention (approximately 2 weeks)
  The investigators will measure participants' anxiety regarding their future career with the Future Career Anxiety Scale. The minimum score is 5 and the maximum is 25. A higher score means a worse outcome (increased anxiety).
Generalised Anxiety symptoms | Change from baseline to post-intervention (approximately 2 weeks)
  The investigators will measure participants' anxiety symptoms using the Generalised Anxiety Disorder Assessment. This is a 7-item instrument that uses the DSM-V criteria to assess anxiety symptom severity. The minimum score is 0 and the highest one is 21. A higher score means a worse outcome (a higher level of anxiety).
Depression symptoms | Change from baseline to post-intervention (approximately 2 weeks)
  The investigators will measure participants' depression symptoms with the Patient Health Questionnaire-9. The scale measures participants' severity of depression using DSM IV criteria. The minimum score is 0 and the highest one is 27. A higher score means a worse outcome (more severe symptoms of depression).
Participants' mental health complaints | Change from baseline to post-intervention (approximately 2 weeks)
  The investigators will measure participants' mental health complaints with the Mental Health Complaints Scale. This is a 5-item instrument that will be used to assess mental health complaints. The minimum score is 6 and the highest is 30. A higher score means a worse outcome.
Participants' psychological capital | Change from baseline to post-intervention (approximately 2 weeks)
  The investigators will measure participants' psychological capital with the 12-item Compound PsyCap Scale. The minimum score is 12 and the highest is 72. A higher score means a better outcome.

OTHER OUTCOMES:
Physical health | Baseline only
  The investigators will use a short version of Ware's Physical Health Complaints Scale to measure participants' perceptions of their health. The minimum score is 4 and the highest is 20. A higher score means a worse outcome (worse physical health).
Treatment adherence | Post-intervention only (approximately 2 weeks)
  Drop out rate; The number of completed assignments; Quality of completed assignment (qualitative rating of the degree of completeness and depth of the answer for each assignment, conducted by two independent experts based on apriori established coding grids).
Satisfaction with the intervention | Post-intervention only (approximately 2 weeks)
  Satisfaction with the intervention will be measured using 17 items. Eleven items are measured on a 4-points, 5-points, and 10-points Likert scale. Each item will be analyzed separately. A higher score means greater satisfaction. The other 6 items are open-ended questions and imply qualitative analysis.
System usability | Post-intervention only (approximately 2 weeks)
  We will use a 10-item questionnaire designed to measure participants' satisfaction with TalentLMS, the online platform used for the program delivery. The total score of System Usability Scale is 0 and the highest one is 100. A higher score means a better outcome.
Sociodemographic information | Baseline only
  Age, gender, residential area, educational level, average monthly income, unemployment period, work experience, and targeted professional field.
Employment status | Follow-up only (approximately 6 weeks)
  Self-reported employment status will be measured at follow-up, using a dichotomous question.
Employment satisfaction | Follow-up only (approximately 6 weeks)
  Self-reported employment quality will be measured at follow-up using 4 questions. One of them is a dichotomous question, while the other 3 questions are measured on a Likert scale. The minimum score is 3, and the maximum is 30. A higher score means greater satisfaction with the job.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Rusu, Principal Investigator — West University of Timisoara
Locations (1):
- West University of Timisoara, Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bangor, A., Kortum, P. & Miller, J. (2009). Determining what individual SUS scores mean: adding an adjective rating scale. Journal of Usability Studies, 4(3), 114-123.
- [Background] Bodnaru, A., Rusu, A., Blonk, R., Vîrgă, D., Iliescu, D., & Van den Broeck, A. (2023, May 4). Bodnaru_et_al_preprint. https://doi.org/10.31234/osf.io/tdseq
- [Background] Blau, G. (1994). Testing a two-dimensional measure of job search behavior. Organizational Behavior and Human Decision Processes, 59, 288-312. https://doi.org/10.1006/obhd.1994.1061
- [Background] Curran, J., Wishart, P., & Gingrich, J. (1999). JOBS: A manual for teaching people successful job search strategies. Ann Arbor: University of Michigan, Institute for Social Research, Michigan Prevention Research Center.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Rosenberg, M. (1979). Conceiving the Self. New York, NY: Basic Books.
- [Background] Saks, A.M., Zikic, J., & Koen, J. (2015). Job search self-efficacy: Reconceptualizing the construct and its measurement. Journal of Vocational Behavior, 86, 104-114. https://doi.org/10.1016/j.jvb.2014.11.007
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Tsai C.T., Hsu H., Hsu Y.C. (2017). Tourism and hospitality college students' career anxiety: Scale development and validation. Journal of Hospitality & Tourism Education, 29(4), 158-165. https://doi.org/10.1080/10963758.2017.1382365
- [Background] Van Hooft, E.A.J., Van Hoye, G., & Van den Hee, S.M. (2022). How to Optimize the Job Search Process: Development and Validation of the Job Search Quality Scale. Journal of Career Assessment, 30(3), 474-505. https://doi.org/10.1177/10690727211052812
- [Background] Virga D, De Witte H, Cifre E. The Role of Perceived Employability, Core Self-Evaluations, and Job Resources on Health and Turnover Intentions. J Psychol. 2017 Oct 3;151(7):632-645. doi: 10.1080/00223980.2017.1372346. Epub 2017 Oct 6. PMID 28985167
- [Background] Vîrga, D. & Rusu, A. (2018). Core self-evaluations, job search behaviour and health complaints. The mediating role of job search self-efficacy. Career Development International, 23(3), 261-273. https://doi.org/10.1108/CDI-11-2017-0208
- [Background] Vuori, J., & Vinokur, A.D. (2005). Job-search preparedness as a mediator of the effects of the Tyohon Job Search Intervention on re-employment and mental health. Journal of Organizational Behavior, 26(3), 275-291. https://doi.org/10.1002/job.308
- [Background] Lorenz T, Beer C, Putz J, Heinitz K. Measuring Psychological Capital: Construction and Validation of the Compound PsyCap Scale (CPC-12). PLoS One. 2016 Apr 1;11(4):e0152892. doi: 10.1371/journal.pone.0152892. eCollection 2016. PMID 27035437
- [Background] Berwick DM, Murphy JM, Goldman PA, Ware JE Jr, Barsky AJ, Weinstein MC. Performance of a five-item mental health screening test. Med Care. 1991 Feb;29(2):169-76. doi: 10.1097/00005650-199102000-00008. PMID 1994148
- [Derived] Bodnaru A, Rusu A, Virga D, Van den Broeck A, Blonk RWB, Tranca LM, Iliescu D. Efficacy of the iJobs Web-Based Psychoeducational Intervention to Improve Job Search Behavior and Promote Mental Health Among Unemployed People: Protocol for a Waitlist Randomized Controlled Trial. JMIR Res Protoc. 2024 May 8;13:e55374. doi: 10.2196/55374. PMID 38717812